CLINICAL TRIAL: NCT05077189
Title: Temporomandibular Joint Complains in Patients With COVID-19
Brief Title: Temporomandibular Joint and COVID-19
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazife Begüm KARAN, Associated Professor, DDS, PhD, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2020/224
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Temporomandibular Disorder; ASA Triad
Keywords: coronavirus; TMJ disorder; DC/TMD; ASA; Sars-CoV-2
MeSH Terms: conditions — COVID-19; Temporomandibular Joint Disorders; Asthma, Nasal Polyps, And Aspirin Intolerance; Coronavirus Infections | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Patients with CV-19 and not in the acute period. This group were then divided into two subgroups each according to ASA (American Society of Anesthesiologist) classification (ASA 1 and ASA 2).
  Interventions: Other: Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) scale
- Control Group: Patients without CV-19 This group were then divided into two subgroups each according to ASA (American Society of Anesthesiologist) classification (ASA 1 and ASA 2).
  Interventions: Other: Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) scale

INTERVENTIONS:
Other: Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) scale — 4 items of the DC/TMD scale were used in this study to evaluate the TMJ disorders.
  1. Demographics Survey
  2. DC/TMD Symptom Questionnaire (SQ)
  3. Graded Chronic Pain Scale (GCPS)
  4. Jaw Functional Limitation Scale-20 (JFLS-20)

SUMMARY:
There is evidence that CV-19 is associated with joint symptoms, but there are no specific data on the temporomandibular joint (TMJ). It is also known that the systemic health status can impact the immune system. Given all this, this study aimed to investigate the effect of CV-19 and systemic health status, as determined by the American Society of Anesthesiologists (ASA) Physical Status Classification System 12, on TMJ in patients with TMJ complaints using the DC/TMD scale.

DETAILED DESCRIPTION:
This study investigates the effect of systemic status, according to American Society of Anesthesiologist (ASA), and COVID-19 on temporomandibular joint (TMJ) disorders using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) scale, shown to be valid for assessing TMJ disorders. The study included 76 patients who presented to our clinic with TMJ. Participants were divided into two groups: those with COVID-19 (CV-19, study group) and those without (non-CV-19, control group). These two groups were both further divided into subgroups according to ASA 1 and ASA 2 classification. Power analyses were performed using G*Power software to determine the required number of patients. Groups were compared using the Symptom Questionnaire, a demographics survey, the Graded Chronic Pain Scale (GCPS), and the Jaw Functional Limitation Scale-20 (JFLS-20) of the DC/TMD. The statistical software program version 1.6.23 was used for statistical analysis. Although joint complaints were more common in ASA 2 patients with CV-19, the groups were not significantly different. The CV-19 ASA 2 group had the highest JFLS-20 score (mean: 1.3±1.5) and the non-CV-19 ASA 1 group had the lowest JFLS-20 score (mean: 0.7±0.8), but the differences were again not significant. Joint complaints were more common and more severe in ASA 2 patients with CV-19, albeit not with statistical significance. More studies are needed to better understand our results.

ELIGIBILITY:
Inclusion Criteria:

* applied to our clinic with TMJ discomfort
* ASA 1 and ASA 2 patients

Exclusion Criteria:

* patients with acute CV-19
* Patients who are not in ASA 1 or ASA 2 classification
* Patients under 18 year-old
* Pregnants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who live in Rize/Turkey
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
DC/TMD scale - Demographics Survey | through study completion an average of 3 months
  This survey consisted of 6 items concerning marital status, socioeconomic status, profession, education, and children.
DC/TMD scale - DC/TMD Symptom Questionnaire | through study completion an average of 3 months
  This 14-item questionnaire aims to determine the duration and causes of pain and the associated symptoms.
DC/TMD scale - Graded Chronic Pain Scale | through study completion an average of 3 months
  This 8-item scale is graded on a scale of 0-10 points. It includes 3 questions on pain intensity, 4 questions on function, and 1 question on the number of days with facial pain. The GCPS consists of two subscales. As the first subscale, Characteristic Pain Intensity is measured, where a score of ≥50 out of 100 possible points indicates high-intensity pain. The Interference Score is then calculated as the second subscale based on scores concerning interference in daily activities and work and the number of days with interference
DC/TMD scale - Jaw Functional Limitation Scale-20 | through study completion an average of 3 months
  This scale consists of three subscales that address limitations of mastication, vertical mobility, and verbal and non-verbal communication. These three subscales are ideal for both research purposes and patient assessment of various functional limitations of the jaw. It is a global scale that consists of 20 items and the three aforementioned subscales (mastication, vertical mobility, and verbal and non-verbal communication)

SECONDARY OUTCOMES:
ASA 1 | through study completion an average of 3 months
  American Society of Anesthesiologist 1 - systemically healthy patients
ASA 2 | through study completion an average of 3 months
  American Society of Anesthesiologist 2 - A patient with mild systemic disease

CONTACTS AND LOCATIONS:
Overall Officials: Nazife B Karan, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Nazife Begüm Karan, Rize, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data that support the other findings in this study are available from the corresponding author upon reasonable request.